CLINICAL TRIAL: NCT04758897
Title: A Dose Ascending, Open Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics Characteristics of VG161 in Subjects With Advanced Malignant Solid Tumors
Brief Title: Clinical Study of VG161 in Subjects With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-C101
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 1. 5.0*10^7 on D1
  2. 1.0*10^8 on D1
  3. 2.0*10^8 on D1
  4. 2.0*10^8 on D1 and D2
  5. 2.0*10^8 on Days 1 to 3
  6. 2.0*10^8 on Days 1 to 4
  7. 2.0*10^8 on Days 1 to 5
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell))

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) — Intratumoral injection only. The dosing date can be the Day 1 only or Days 1 through 5.
  Other Names: VG161

SUMMARY:
VG161 is a recombinant human-IL12/15/PDL1B oncolytic HSV-1 Injectable. This Phase I study will be conducted in HSV-seropositive subjects with advanced malignant solid tumors that are refractory to conventional therapies. This is an open label study to determine the safety and tolerability of VG161, and recommended dose of VG161 for Phase II trials.

DETAILED DESCRIPTION:
The trial will be conducted in 7 dose ascending cohorts, including 3 single dose accelerated titration design pilots and 4 multiple dose escalation groups.

Descriptive statistics will be used to summarize all data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged within 18 to 80 years.
2. Subject with late stage carcinoma which is refractory/relapsed after and/or intolerant of standard therapies or for which no standard therapy exists.
3. There is at lease one injectable tumor lesion that meet the requirements of the assigned dose level. The superficial lesions are preferred, and the deep lesions that can be injected under the guidance of B ultrasound or computed tomography (CT) scan can also be selected.
4. Eastern Cooperative Oncology Group (ECOG) scores 0 or 1.
5. Life expectancy is at least 3 months.
6. Required organ function:

1) Hematology blood (no blood transfusion or colony stimulating factor treatment within 14 days): Absolute neutrophil count (ANC)≥1.5×10^9L, Platelets ( PLT)≥75×10^9L, hemoglobin (Hb)≥85g/L; 2) Liver function: Total Serum bilirubin (TBIL)≤1.5×ULN (the upper limit of the reference range), Alanine aminotransferase (ALT)≤3×ULN, aspartate aminotransferase (AST)≤3×ULN (acceptable for patients with liver metastasis or liver cancer: TBIL≤5×ULN, AST≤5×ULN, ALT≤5×ULN); 3) Renal function: Serum creatinine≤1.5×ULN, and creatinine clearance≥50 ml/min (calculated per Cockcroft-Gault formula); 4) Coagulation function: activated partial thromboplastin time (APTT)≤1.5×ULN, international standardized ratio (INR)≤1.5×ULN.

7. Subjects of childbearing potential (male and female) must agree to use a reliable contraceptive method (hormone or barrier method or abstinence) during the study and for at least 90 days following the last dose; females of childbearing potential must have a negative blood or urine pregnancy test within 7 days of study enrollment.

8. Signed written informed consent.

Exclusion Criteria:

1. Subject in prior anti-tumor therapies such as chemotherapy, radiotherapy, biotherapy, endocrinotherapy, targeted therapy, immunotherapy within 4 weeks of study treatment initiation.
2. Participation in clinical trials of any other investigational agents within 4 weeks of study treatment initiation.
3. Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks of study treatment initiation.
4. Patients who received systemic treatment with either corticosteroids ( >10 mg/ daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study treatment initiation.
5. Subjects with any ≥Grade 1 toxicity (as per NCI CTC AE Version 5.0) related to prior anti-cancer therapy (except for toxicity that the investigator assessed to be no safety risk, such as alopecia.).
6. Subjects with any uncontrolled active Central Nervous System (CNS) metastasis or meningeal metastasis with clinical symptoms.
7. Seronegative for Herpes Simplex Virus (HSV) (HSV-1IgG and HSV-1IgM).
8. Subjects with the relapse of HSV infection and relevant clinical manifestations, such as lip herpes, herpes keratitis, herpes dermatitis, and genital herpes.
9. Subjects with other uncontrolled active infections.
10. Known history of immunodeficiency and test positive of human immunodeficiency virus (HIV).
11. Active infection of hepatitis B (HBV) (hepatitis b virus titer higher than the detection limit or those requiring antiviral therapy), or hepatitis C virus (HCV).
12. History of severe cardiovascular disease:

1)Ventricular arrhythmias requiring clinical intervention; 2)QTc interval >480 ms; 3)Acute coronary syndrome, congestive heart failure, stroke or other cardiovascular events of III grade or above within 6 months; 4)The cardiac function grade≥II or left ventricular ejection fraction (LVEF) <50% per the New York Heart Association (NYA); 5)Uncontrolled hypertension. 13. Subjects with active or past autoimmune diseases that are likely to recur (e.g. systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); acceptable for patients with clinically stable autoimmune thyroiditis.

14. Subjects with any prior ≥Grade 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent.

15. known to have alcohol or drug dependence. 16. Persons with mental disorders or poor compliance. 17. Pregnant or lactating women. 18. Subjects with any significant unrelated systemic illness that to the investigator's opinion would compromise the subject's eligibility to participate the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-03-14 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
MTD/RP2D | 1 month
  MTD (Maximum tolerable dose) / RP2D (Recommended dose for phase II)
Occurence of DLT | 1 month
  Occurence of DLT (Dose Limiting Toxicity)
Numbers of DLT | 1 month
  Numbers of DLT (Dose Limiting Toxicity)
Occurence of AE and SAE（NCI CTCAE 5.0） | 7 months
  Occurence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Frequency of AE and SAE（NCI CTCAE 5.0） | 7 months
  Frequency of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）

SECONDARY OUTCOMES:
Tmax(h) | At the end of Cycle 1 (each cycle is 28 days)
  Time to peak
Cmax(copies/ugDNA) | At the end of Cycle 1 (each cycle is 28 days)
  Maximum concentration
ORR | 7 months
  Evaluate Objective Response Rate by RECIST 1.1.
DCR | 7 months
  Evaluate Disease Control Rate by RECIST 1.1.
mPFS | 7 months
  Evaluate medium Progression Free Survival by RECIST 1.1.
CD3+, CD4+, CD8+ | 7 months
  Concentration of CD3+, CD4+, CD8+
IL15 | 7 months
  Concentration of IL15
PD-L1, PD-1 | 7 months
  Concentration of PD-L1, PD-1,
Existence of Biomarkers | 4 months
  PD-L1, Nectin2, HVEM

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, doctor, Principal Investigator — Shanghai East Hospital
Locations (2):
- China (2):
  - ShangHai East hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to ShangHai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No